CLINICAL TRIAL: NCT00258921
Title: An International Registry in Essential Hypertension
Brief Title: RIAT Registry: Reason for Not Intensifying Antihypertensive Treatment
Acronym: RIAT
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Other Study IDs: R-9511
Record Dates: First submitted 2005-11-24; First posted 2005-11-28 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2007-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
To support physicians in their active management of hypertensive patients. By targeting specific systolic and diastolic blood pressure (BP) figures physicians will closely monitor the BP values and as such will have an individualized control of the treatment in each patient.

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

Main criteria are listed hereafter:

Inclusion Criteria:

* Adult hypertensive
* Either newly diagnosed and untreated
* or previously treated and uncontrolled Patients of both sexes with essential hypertension

Exclusion Criteria:

* Known secondary hypertension
* Known secondary curable hypertension (i.e. pheochromocytoma, aldosterone producing adenoma, Cushing disease). Patients with renal disease are not excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31870
Dates: Start 2004-03; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pascale BLONDIN, MD, Study Director — Sanofi